CLINICAL TRIAL: NCT07375082
Title: Rehabilitation Approaches Used by Physiotherapists Following Total Knee Replacement- a Cross-sectional Survey
Brief Title: Rehabilitation Approaches Used in Total Knee Replacement
Status: Active, not recruiting | Type: Observational
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Rabia Khan, Assistant Professor, Bahria University
Other Study IDs: BUHS-IRB # 225/25
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Osteo Arthritis of the Knee; Rhematoid Arthritis
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnare will be filled by physiotherpist

SUMMARY:
In this study, we will investigate the rehabilitation approaches commonly used by physiotherapists in Pakistan following total knee replacement. Total knee replacement is a frequently performed surgical procedure, and effective postoperative rehabilitation is essential for improving pain, mobility, and functional outcomes.

A web-based cross-sectional survey will be conducted among practicing physiotherapists from different provinces of Pakistan. Data will be collected using a structured questionnaire to explore demographic characteristics, rehabilitation techniques employed at various stages of recovery, and challenges faced in post-TKR rehabilitation. The collected data will be analyzed using appropriate descriptive and inferential statistical methods.

The findings will help identify prevailing rehabilitation practices and variations among physiotherapists. This study will contribute to understanding current clinical trends, identifying gaps in practice, and promoting the use of evidence-based and standardized rehabilitation protocols. Ultimately, the results will support improved patient recovery, guide professional training, and assist in developing consistent post-TKR rehabilitation strategies in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Currently practicing physiotherapists of Pakistan
* clinical experience more than 5 years

Exclusion Criteria:

* Physiotherapists have clinical experience less than 5 years
* Academic Physiotherapist only

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of practicing physiotherapists in Pakistan who are actively involved in clinical rehabilitation. Participants will be recruited from various provinces, including Punjab, Sindh, Khyber Pakhtunkhwa, Balochistan, and the Islamabad Capital Territory. Physiotherapists working in diverse healthcare settings such as public and private hospitals, rehabilitation centers, orthopedic clinics, and outpatient departments will be included to ensure broad representation.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
determine the type of rehabilitation approaches | 3 months
  This observational study will document and classify the type of post-operative rehabilitation received by patients following Total Knee Replacement (TKR) over a 3-month (12-week) period using a structured questionnaire, without assigning or altering treatment

SECONDARY OUTCOMES:
identify variations in rehabilitation practices | 3 months
  Rehabilitation practices after Total Knee Replacement vary widely during the first 3 months post-surgery with respect to setting (inpatient facility, outpatient clinic, home, or community), level of supervision (fully supervised, remotely supervised, or unsupervised), mode of delivery (individual, group-based, or telerehabilitation), and rehabilitation dose (timing of initiation, session frequency, duration, and total number of sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Khan, Masters of Science, Principal Investigator — Bharia University Health Sciences Campus Karachi
Locations (1):
- Bahria University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Sekamova SM, Beketova TP. [Morphological bases of liver insufficiency in the early stages of the prolonged crush syndrome]. Biull Eksp Biol Med. 1985 Nov;100(11):614-7. Russian. PMID 4063514